CLINICAL TRIAL: NCT06493058
Title: Evaluatıon of the Effectiveness of the Prone Position in Babies Extubed After Congenital Cardio Surgery
Brief Title: Extruded the effectıveness of Prone posıtıon ın ınfants evaluatıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-3150
Record Dates: First submitted 2024-04-20; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Prone posıtıon
Keywords: Congenital Heart Diseases; Extubation; Newborn; Prone Position
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Prone Position

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In our study, the babies in the study group were given the supine, right lateral and left lateral positions (12×1), which are used in nursing care practices in the clinic after extubation, in addition to the supine, right lateral and left lateral positions (12×1), the prone position was given twice a day for 2×2 hours twice a day within 48 hours after extubation, with the head on the midline of the neck and the head facing to the right or left side.
  Interventions: Other: Prone positioning
- Control group (No Intervention): Babies in the control group did not receive any treatment.

INTERVENTIONS:
Other: Prone positioning — The babies in the study group were given the supine, right lateral and left lateral positions (12×1), which are used in nursing care practices in the clinic after extubation, in addition to the supine, right lateral and left lateral positions (12×1), the prone position was given twice a day for 2×2 hours twice a day within 48 hours after extubation, with the head on the midline of the neck and the head facing to the right or left side.
  Arms: Intervention group

SUMMARY:
The aim of this study was to determine the effect of prone position on vital signs, arterial blood gases and blood values in 0-1 year old infants extubated after congenital heart surgery. The study was a randomised controlled experimental type study.

DETAILED DESCRIPTION:
The sample of the study consisted of 40 infants aged 0-1 year who underwent surgery in the Cardiovascular Surgery Intensive Care Unit of a private hospital.Data collection tools consisted of "Data Collection Form", "Vital Signs Follow-up Form", "Arterial Blood Gas Follow-up Form", "Blood Values Follow-up Form" prepared by the researcher in line with the literature information and some measurement data used in the study (arterial blood sample obtained with the blood gas measurement device used in the NICU and blood gas parameters (PaCO2, pH, PaO2, Lac and SaO2) and bedside monitor).

The study was conducted in the Cardiovascular Surgery Intensive Care Unit of a private foundation university hospital. Infants between the ages of 0 and 1 year who had undergone congenital heart surgery and were extubated after surgery, who did not have any congenital anomalies of the lungs in addition to congenital heart disease, who did not have any condition that could affect cardiac, circulatory and respiratory functions or prevent positioning were included in the study. The infants to be included in the study were randomly selected to the control and study groups to avoid bias in the study. Which of the experimental or control groups the infants included in the study would be in was determined by using the address "https://www.calculatorsoup.com".

ELIGIBILITY:
Inclusion Criteria:

* To be between 0-1 years old
* Having congenital heart surgery
* Endotracheal intubation has been applied
* Being extubated after congenital heart surgery
* Obtaining permission from their parents to participate in the study

Exclusion Criteria:

* In addition to the diagnosis of congenital heart disease, congenital heart disease of the lungs with any of the anomalies,
* Position that may affect cardiac, circulatory and respiratory functions or surgical intervention that prevents ECMO (open sternum bone, ECMO support, etc.)
* Complications developed during the study,
* Infants whose parents did not agree to participate in the study were included in the study. is not recognised.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Life Findings Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  Pulse values were monitored for 48 hours
Life Findings Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  Saturation values were monitored for 48 hours
Life Findings Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  Blood pressure values were monitored for 48 hours

SECONDARY OUTCOMES:
Arterial Blood Gas Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  After positioning, potansiyel hidrojen in blood were evaluated.
Arterial Blood Gas Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  After positioning, Partial arterial oxygen pressure, were evaluated.
Arterial Blood Gas Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  After positioning, Partial arterial carbon dioxide pressure were evaluated.
Arterial Blood Gas Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  After positioning, Arterial oxygen saturation were evaluated.
Arterial Blood Gas Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  After positioning, Laktat, were evaluated.
Arterial Blood Gas Monitoring Form | Taken immediately before extubation and at 8, 16, 24, 32 and 48 hours after extubation
  After positioning, arterial blood gases were evaluated.

OTHER OUTCOMES:
Blood Values Monitoring Form | Ekstübasyondan hemen önce ve ekstübasyon sonrası 24. ve 48. saatlerde alındı
  Hemoglobin were evaluated.
Blood Values Monitoring Form | Taken immediately before extubation and at 24 and 48 hours after extubation
  Hematocrit were evaluated.
Blood Values Monitoring Form | Taken immediately before extubation and at 24 and 48 hours after extubation
  Leukocyte were evaluated.
Blood Values Monitoring Form | Taken immediately before extubation and at 24 and 48 hours after extubation
  Platelet were evaluated.
Blood Values Monitoring Form | Taken immediately before extubation and at 24 and 48 hours after extubation
  Procalcitonin were evaluated.
Blood Values Monitoring Form | Taken immediately before extubation and at 24 and 48 hours after extubation
  C-reaktif protein were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kökcü Doğan, Study Director — Istanbul Meidpol University
Locations (1):
- Istanbul Meidpol University Hospital, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No